CLINICAL TRIAL: NCT00231192
Title: Repaglinide for Adolescents With Cystic Fibrosis-Related Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit any subjects
Sponsor: Children's Hospital of Philadelphia (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-8-4323; Cystic Fibrosis Foundation
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2007-11

CONDITIONS: Diabetes
Keywords: Diabetes; Adolescents; Cystic Fibrosis; Insulin; Repaglinide
MeSH Terms: conditions — Diabetes Mellitus; Cystic Fibrosis; Insulin Resistance | interventions — repaglinide; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Repaglinide and Insulin

SUMMARY:
This study will test the hypothesis that oral repaglinide is equivalent to insulin in the treatment of new-onset CFRD in adolescents. In addition, successful treatment of CFRD with repaglinide will improve nutritional status, ameliorate declines in pulmonary function, and will not have a negative impact upon quality of life.

DETAILED DESCRIPTION:
This study will test the hypothesis that oral repaglinide is equivalent to insulin in the treatment of new-onset CFRD. This hypothesis will be tested using the following aims:

Specific Aim 1: To determine the effect of three months of repaglinide and insulin treatment upon blood glucose (BG) and insulin excursion during an oral glucose tolerance test.

Specific Aim 2: To determine the effect of three months of repaglinide and insulin treatment upon BG as measured by continuous glucose monitoring, fasting BG, 2-hour post-prandial BG, hemoglobin A1C, and serum fructosamine.

Secondary Aim 1: To determine the effect of three months of repaglinide and insulin treatment upon weight, body mass index, and lean body mass in adolescents with new-onset CFRD.

Secondary Aim 2: To determine the effect of three months of repaglinide and insulin treatment upon pulmonary function in adolescents with new-onset CFRD.

Secondary Aim 3: To determine the effect of three months of repaglinide and insulin treatment upon quality of life in new-onset CFRD.

ELIGIBILITY:
Inclusion Criteria:

Cystic Fibrosis, Blood glucose concerning for diabetes -

Exclusion Criteria:

Known Cystic Fibrosis-Related Diabetes, Liver Disease, FEV1<40%

-

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2005-10; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
blood glucose
insulin excursion during oral glucose tolerance test
fasting blood glucose
2-hour post-prandial blood glucose
hemoglobin A1C
serum fructosamine

SECONDARY OUTCOMES:
weight
body mass index
lean body mass
pulmonary function
quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kelly, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States